CLINICAL TRIAL: NCT05042700
Title: The Effect of Melatonin in Patients With Low Anterior Resection Syndrome
Acronym: MELLARS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ismail Gögenur (Other)
Collaborators: Hvidovre University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Ismail Gögenur, Professor, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REG-140-2020; 2020-004442-11 (EudraCT Number)
Record Dates: First submitted 2021-08-30; First posted 2021-09-13 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Low Anterior Resection Syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin-Placebo sequence (Experimental): 50% of the included patients will receive 4 weeks of treatment with melatonin, followed by a 4 week wash out period, and then 4 weeks of treatment with placebo. The treatments are blinded.
  Interventions: Drug: Melatonin; Drug: Placebo
- Placebo-Melatonin sequence (Experimental): 50% of the included patients will receive 4 weeks of treatment with placebo, followed by a 4 week wash out period, and then 4 weeks of treatment with melatonin. The treatments are blinded.
  Interventions: Drug: Melatonin; Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Enema with 25 mg melatonin
Drug: Placebo — Enema without melatonin

SUMMARY:
The primary objective of the study is to investigate whether treatment with melatonin has an alleviating effect on Low Anterior Resection Syndrome (LARS) symptoms. Secondarily, the effect of the treatment on bowel movements, other patient reported symptoms, quality of life, depression, anxiety, sleep disturbances, motilin levels, and microscopic changes in rectal mucosa will be investigated.

DETAILED DESCRIPTION:
This trial which will be conducted in two phases.

The first part of the study will be conducted as an internal feasibility test. Three patients with major LARS will be included. Patients will be recruited from the Department of Surgery, Zealand University Hospital. These patients will not be randomized nor blinded. They will receive a 4-week treatment with 25 mg melatonin and will undergo the same questionnaires and tests before and after treatment as in the randomized clinical trial. The preliminary results from the internal feasibility test will allow us to assess potential difficulties related to the administration or design, which then will be able to be corrected before the randomization part is initiated.

The second part of the will be conducted as a randomized, blinded, placebo-controlled, crossover study and will be testing whether treatment with melatonin has an alleviating effect on Low Anterior Resection Syndrome (LARS) symptoms.

Patients will be randomized to receive 4 weeks of treatment with melatonin, followed by a 4 week wash out period, and then 4 weeks of treatment with placebo (M-P) or 4 weeks of treatment with placebo, followed by a 4 week wash out period, and then 4 weeks of treatment with melatonin (P-M). Both participants and investigators will be blinded.

Patients will be given questionnaires before and after each treatment period to assess outcomes. Blood samples and rectal biopsies will be taken after each treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should have major LARS (LARS score >29).
2. Patients should have undergone bowel continuity restoring surgery between the last 3 to 24 months.
3. Participants should be 18 years or older.
4. Participants must sign an informed consent form.

Exclusion Criteria:

1. Known allergic reaction to melatonin.
2. Dementia as determined by mini mental state examination score (MMSE) < 24.
3. Participation in another pharmacological intervention trial at the point of inclusion.
4. Completed any adjuvant oncological treatment within the last three months.
5. Ongoing oncological treatment.
6. Rotor or Dubin-Johnson syndrome, epilepsy, systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), Parkinson's disease, spinal cord injury and multiple sclerosis.
7. Severe liver disease defined as transaminases above 3 times the normal levels, and severe kidney disease defined as eGFR below 40 ml/min.
8. Daily ongoing hypnotic treatment.
9. Pre-existing medical sleep disorder diagnosed before the diagnosis of rectal cancer (i.e sleep apnea, restless legs, narcolepsy.)
10. Work involving nightshifts.
11. Daily alcohol consumption above 5 units of alcohol (1 unit = 12 g alcohol)
12. Predictable poor compliance (due to pre-existing psychiatric disease, dementia or not able to read or speak sufficient Danish)
13. Pregnant or breastfeeding.
14. Severe, life-threatening medical condition, that implies that the patient cannot participate in the study course. (e.g. metastatic disease, local recurrence, stroke, AMI).
15. Females not in menopause (defined as no menstruation during the last 12 months) should not be pregnant. Furthermore, reproductive females should use a secure birth control (intrauterine devices, hormonal contraceptives including - oral pills, patches, vaginal rings and injections) during the entire period of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Low Anterior Resection Syndrome Score | 4 weeks
  The LARS Score questionnaire is filled out by the participants before and after each treatment period.

SECONDARY OUTCOMES:
Daily bowel function | 4 weeks
  The participants will fill out a diary on the daily bowel movements during the treatment phase
Self-reported quality of life | 4 weeks
  EORTC Quality of Life Questionnaire for cancer patients and specifically colorectal cancer patients
Other patient reported symptoms | 4 weeks
  Measure Yourself Medical Outcome Profile (MYMOP) is a self-administered questionnaire. Patients are asked to specify one or two symptoms that concern them the most. Subsequently they evaluate the severity on a 7-point Likert scale. The second part of the questionnaire uses the same scale to assess whether the symptom limits or prevent any daily activity, and also to rate general well-being. Follow-up questionnaires address the original issues completed in the initial form. Symptom 1, symptom 2, activity, and wellbeing each have a separate score between 0 and 6 with 0 indicating "as good as it could be" and 6 "as bad as it could be". An overall score is calculated by taking the average of item scores.
Anxiety | 4 weeks
  Hospital Anxiety and Depression Scale (HADS-A): The anxiety subscale consists of 7 questions which are graded on a 4 point scale (0-1-2-3) and is summed into a total score between 0-21. A score of 7 or lower is negative case, a score of 8 - 10 is a doubtful case, and a score of 11 or above is a positive case.
Depression | 4 weeks
  Hospital Anxiety and Depression Scale (HADS-D): The depression subscale consists of 7 questions which are graded on a 4 point scale (0-1-2-3) and is summed into a total score between 0-21. A score of 7 or lower is negative case, a score of 8 - 10 is a doubtful case, and a score of 11 or above is a positive case.
Sleep | 4 weeks
  Participants will wear an actigraph during the treatment phases and fill out a sleep diary and this will allow to asses sleep time (minutes).
Insomnia | 4 weeks
  Insomnia Severity Index (ISI)
Incidence of treatment-emergent Adverse Effects [Safety and reactions] | 4 weeks
  Participants will be systematically interviewed before and after the treatment periods.
Melatonin | 4 weeks
  Blood samples will be taken after each treatment ends.
Multiplex gene assay - NanoString nCounter® Inflammation Panel analysis in blood | 4 weeks
  Difference in gene expressions between intervention and placebo groups
Motilin | 4 weeks
  Blood samples will be taken after each treatment ends.
Pathological assessment of inflammation | 4 weeks
  Rectal biopsies will be taken after each treatment ends.The FFPE treated biopsies will be assessed by pathologist using a routine inflammatory grading system to asses inflammation
Multiplex gene assay - NanoString nCounter® Inflammation Panel analysis in biopsies | 4 weeks
  Difference in gene expressions between intervention and placebo groups
Motilin receptors | 4 weeks
  Rectal biopsies will be taken after each treatment ends.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, DMSc, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zahid JA, Madsen MT, Bulut O, Christensen P, Gogenur I. Effect of melatonin in patients with low anterior resection syndrome (MELLARS): a study protocol for a randomised, placebo-controlled, crossover trial. BMJ Open. 2023 Sep 11;13(9):e067763. doi: 10.1136/bmjopen-2022-067763. PMID 37696629